CLINICAL TRIAL: NCT01708707
Title: A Randomized Comparison of Sublingual Buprenorphine to Morphine Sulfate in the Treatment of Neonatal Abstinence Syndrome (NAS)
Brief Title: Comparison of Buprenorphine to Morphine in Treatment of Neonatal Abstinence Syndrome (NAS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pediatrix (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Banner IRB 01-13-0030
Record Dates: First submitted 2012-04-25; First posted 2012-10-17 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-03

CONDITIONS: Neonatal Abstinence Syndrome; Neonatal Withdrawal Syndrome
MeSH Terms: conditions — Neonatal Abstinence Syndrome | interventions — Buprenorphine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral morphine sulfate (Active Comparator): Oral morphine sulfate 0.4 mg/kg/day morphine every 3-4 hours as needed for Finnegan scores suggestive of Neonatal Abstinence Syndrome Other Name: morphine
  Interventions: Drug: Morphine Sulfate
- Buprenorphine (Experimental): Sublingual Buprenorphine 15.9 µg/kg per day in 3 divided doses, titrated up or escalated down based upon standardized scoring for neonatal abstinence syndrome
  Interventions: Drug: Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine — The injectable formulation of buprenorphine (Buprenex; Reckitt Benckiser) will be prepared to a final concentration of 0.075 mg/mL in 100% ethanol and simple syrup USP to create a sublingual preparation.
  Infants initial dose: 15.9 µg/kg per day in 3 divided doses with escalation/weaning based upon standardized scoring of NAS symptoms, using standardized Finnegan scoring Maximum dosage: 60 µg/kg per day Duration: Infants will receive buprenorphine until they are successfully weaned off of opioids and no longer show withdrawal symptoms, evidenced by low Finnegan scores. Mean use in other investigations was 24 days.
  Other Names: Sublingual buprenorphine; Other Name: Buprenex (buprenorphine); NDC Number: 12496-0757-1; Product Code: 12496-0757
  Arms: Buprenorphine
Drug: Morphine Sulfate — Oral Morphine Sulfate Dosage: Morphine Sulfate Oral Solution 100mg/5mL Initially dosed at 0.4mg/kg per day in six daily doses Duration of medication administration dependent upon infant symptoms of neonatal withdrawal, with mean duration of use at Banner Good Samaritan Hospital currently averaging 25 days.
  Other Names: Oral Morphine Sulfate; Morphine; NDC: 0406-8003-24
  Arms: Oral morphine sulfate

SUMMARY:
The purpose of the study is to determine whether buprenorphine is a beneficial, safe, cost effective treatment alternative to morphine sulfate in the treatment of Neonatal Abstinence Syndrome (NAS).

DETAILED DESCRIPTION:
Neonatal abstinence syndrome is a condition that affects newborns who are exposed to chronic opioid drugs while they are in a mother's uterus (womb) prior to birth. The current standard of care treatment includes morphine sulfate. Buprenorphine is a drug used in adults to treat narcotic dependence and withdrawal, but has not yet been approved for use in newborns as a treatment alternative for Neonatal Abstinence Syndrome. This investigation is designed to measure if sublingual (under the tongue) buprenorphine is able to reduce hospital length of stay and decrease number of days of drug treatment currently required in treatment of NAS. Another goal will be to understand buprenorphine as a cost effective treatment for NAS.

ELIGIBILITY:
Inclusion Criteria:

* Infants of corrected gestational age ≥37 weeks
* Chronic opioid exposure in utero
* Signs and symptoms of NAS requiring treatment
* 2 consecutive Finnegan scores ≥8 or any single score ≥12

Exclusion Criteria:

* Concomitant maternal benzodiazepine or alcohol use 30 days prior to enrollment
* Life-threatening congenital malformations
* Intrauterine growth retardation
* Seizure activity or congenital neurologic abnormalities
* Concomitant neonatal use of Cytochrome P450 inhibitor or inducers prior to treatment
* Inability of mother's consent due to altered mental status or comorbid psychiatric disorder
* Neonatal administration of morphine prior to enrollment into study

Max Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2012-12; Primary Completion 2017-10 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | Up to hospital discharge, an anticipated average of 4 weeks
  Number of days of hospital admission

SECONDARY OUTCOMES:
Number of adverse or serious adverse events | Up to hospital discharge, with length of stay currently averaging approximately 4 weeks
Cost efficiency of buprenorphine | At least 48 prior to hospital discharge, with anticipated discharge averaging to be 4 weeks
  Cost of buprenorphine as a product of number of days of administration
Withdrawal symptoms | Up to hospital discharge, usually occuring on average 4 weeks
  Finnegan methodology to score withdrawal symptoms every four hours of medication administration
Rescue dosage administration | Up to hospital discharge, anticipating an average of 4 weeks
  Number of rescue doses of additional medication

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Martin, MD, Principal Investigator — Banner University Medical Center
Locations (1):
- Banner - University Medical Center Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Zankl A, Martin J, Davey JG, Osborn DA. Opioid treatment for opioid withdrawal in newborn infants. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD002059. doi: 10.1002/14651858.CD002059.pub4. PMID 34231914